CLINICAL TRIAL: NCT00140751
Title: A 48-Weeks National Multicenter Randomized Open Clinical Trial Evaluating Tolerance and Efficacy of a Treatment Simplification by Lopinavir/Ritonavir Versus Continuation of Current Treatment in HIV-Infected Patients With a Viral Load Inferior to 50 Copies/mL Since 6 Months At Least
Brief Title: Comparison of Treatment Simplification by LPV/r vs Current Treatment Continuation in HIV-Infected Patients
Acronym: KALESOLO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institut de Médecine et d'Epidémiologie Appliquée - Fondation Internationale Léon M'Ba (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMEA-030; KALESOLO
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2013-09-19 (Estimated); Status verified 2013-09

CONDITIONS: HIV Infections
Keywords: HIV-1; Treatment simplification; Lopinavir/ritonavir; Treatment Experienced; HIV Seropositivity
MeSH Terms: conditions — HIV Infections; HIV Seropositivity | interventions — Lopinavir; Ritonavir; Pharmaceutical Preparations

ARMS (2):
- Simplification (Experimental): The patients included in this arm are on Monotherapy of Kaletra (Lopinavir/ritonavir)during 48 weeks
  Interventions: Drug: Lopinavir/ritonavir (drug)
- Continued (No Intervention): The patients included in this arm continue their treatment without any changes

INTERVENTIONS:
Drug: Lopinavir/ritonavir (drug)
  Arms: Simplification

SUMMARY:
The purpose of this study is to compare the efficacy and tolerance of a treatment simplification by a Lopinavir/ritonavir monotherapy versus continuation of current treatment in HIV-infected patients

DETAILED DESCRIPTION:
Highly active antiretroviral therapy (HAART) has made a significant impact on the natural history of HIV-1 infection, but toxicities and complexities of therapy limit long-term efficacy, and make simpler yet effective HAART regimens highly desirable. Previous attempts to 'de-intensify' protease inhibitor (PI)-based therapy by discontinuing reverse transcriptase inhibitors (RTI) after achieving viral suppression met with failure, probably because plasma levels of most individually administered PI are too low to inhibit viral replication consistently.

Low-dose ritonavir substantially enhances lopinavir plasma levels, and lopinavir/ritonavir (LPV/r) is effective as part of a combination therapy in both naive and PI-experienced patients. Furthermore, lopinavir is known to have a high genetic barrier to selection of resistance. LPV/r monotherapy could thus have the right combination of potency, favorable pharmacokinetics, and high genetic barrier needed to suppress viral replication and prevent the selection of lopinavir resistance. Preliminary results with "maintenance"LPV/r monotherapy show interesting results but data from randomized studies are needed.

ELIGIBILITY:
Inclusion Criteria:

* Age > or = 18 years
* Confirmed HIV-1 seropositivity
* Antiretroviral treatment stable since 3 months at least
* HIV-1 ARN load < 50 copies/mL since 6 months at least
* Signed consent form
* No history of treatment failure (= viral load > 1000 copies/mL) including a protease inhibitor
* No opportunistic infection in the previous 6 months

Exclusion Criteria:

* Neutrophils < 750/mm3
* Hemoglobin < 8 g/dL
* Platelets < 60,000/mm3
* Creatinin > 150 micromoles/L
* SGOT > 5 NUL (Normal Upper Limit)
* SGPT > 5 NUL
* Current IL-2 treatment
* HBV infection treated or not by lamivudine or tenofovir
* Pregnancy or feeding
* Enrollment in another study not compliant with KALESOLO Study group assignment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2005-10; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with a viral load < 50 copies/mL at S48 without any modification of antiretroviral treatment during study | W48

SECONDARY OUTCOMES:
Durability of viral response | W48
Evolution of lymphocytes CD4 | W48
Observance | W48
Clinical and biological tolerance | W48
Quantitative and qualitative changes in quality of life data | W48
Cost-efficacy ratio | W48
Predictive value of proviral DNA before treatment simplification | W48
Proportion of patients showing a lipodystrophy at J0 and S48 | W48

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc MEYNARD, MD, PhD, Principal Investigator — Hôpital Saint-Antoine - Service des Maladies Infectieuses et Tropicales (Paris, France)
Locations (25):
- France (25):
  - Hôpital Pierre Zobda-Quitman - Service de Maladies Infectieuses et Tropicales, Fort-de-France, Martinique
  - Centre Hospitalier de la Région Annecienne (CHRA) - Service d'Infectiologie, Annecy
  - Hôpital Jean Verdier - Unité de Maladies Infectieuses, Bondy
  - Hôpital Pellegrin - Service de Médecine Interne et Maladies Infectieuses, Bordeaux
  - Hôpital Saint-André - Service de Médecine Interne et Maladies Infectieuses, Bordeaux
  - Hôpital Saint-André - Service de Médecine Interne et Maladies Tropicales, Bordeaux
  - Hôpital Côte de Nacre - Service des Maladies Infectieuses, Caen
  - Hôpital Henri Mondor - Service d'Immunologie Clinique, Créteil
  - Hôpital Raymond Poincaré - Service des Maladies Infectieuses et Tropicales, Garches
  - Hôpital A. Michallon - Service des Maladies Infectieuses, Grenoble
  - Hôpital Bicêtre - Service de Médecine Interne, Le Kremlin-Bicêtre
  - Hôpital Nord - CISIH, Marseille
  - Hôpital Sainte-Marguerite - Unité Médicale CISIH, Marseille
  - Hôpital Gui de Chauliac - Service de Maladies Infectieuses et Tropicales, Montpellier
  - Hôpital de l'Archet - Service d'Infectiologie, Nice
  - Hôpital Saint-Antoine - Service des Maladies Infectieuses et Tropicales, Paris
  - Groupe Hospitalier Pitié-Salpêtrière - Service de Maladies Infectieuses et Tropicales, Paris
  - Groupe Hospitalier Pitié-Salpêtrière - Service de Médecine Interne 1, Paris
  - Hôpital-Fondation Saint-Joseph - Service des Maladies Infectieuses, Paris
  - Hôpital Européen Georges Pompidou (HEGP) - Département d'Immunologie, Paris
  - Hôpital Tenon - Service des Maladies Infectieuses et Tropicales, Paris
  - Hôpital Pontchaillou - Service des Maladies Infectieuses, Rennes
  - Hôpital Civil - Hôpital de Jour du CISIH - Clinique Médicale A, Strasbourg
  - Hôpital Gustave Dron - Service des Maladies Infectieuses, Tourcoing
  - Hôpital de Brabois Adultes - Service de Maladies Infectieuses et Tropicales, Vandœuvre-lès-Nancy

REFERENCES:
- [Background] Mocroft A, Ledergerber B, Katlama C, Kirk O, Reiss P, d'Arminio Monforte A, Knysz B, Dietrich M, Phillips AN, Lundgren JD; EuroSIDA study group. Decline in the AIDS and death rates in the EuroSIDA study: an observational study. Lancet. 2003 Jul 5;362(9377):22-9. doi: 10.1016/s0140-6736(03)13802-0. PMID 12853195
- [Background] Yeni PG, Hammer SM, Hirsch MS, Saag MS, Schechter M, Carpenter CC, Fischl MA, Gatell JM, Gazzard BG, Jacobsen DM, Katzenstein DA, Montaner JS, Richman DD, Schooley RT, Thompson MA, Vella S, Volberding PA. Treatment for adult HIV infection: 2004 recommendations of the International AIDS Society-USA Panel. JAMA. 2004 Jul 14;292(2):251-65. doi: 10.1001/jama.292.2.251. PMID 15249575
- [Background] Bartlett JA, DeMasi R, Quinn J, Moxham C, Rousseau F. Overview of the effectiveness of triple combination therapy in antiretroviral-naive HIV-1 infected adults. AIDS. 2001 Jul 27;15(11):1369-77. doi: 10.1097/00002030-200107270-00006. PMID 11504958
- [Background] Palella FJ Jr, Delaney KM, Moorman AC, Loveless MO, Fuhrer J, Satten GA, Aschman DJ, Holmberg SD. Declining morbidity and mortality among patients with advanced human immunodeficiency virus infection. HIV Outpatient Study Investigators. N Engl J Med. 1998 Mar 26;338(13):853-60. doi: 10.1056/NEJM199803263381301. PMID 9516219
- [Background] Murphy R, Gazzard B. Antiretroviral treatment guidelines. AIDS. 2003 Jun;17 Suppl 2:S1. doi: 10.1097/00002030-200306002-00001. No abstract available. PMID 12870522
- [Background] Bucher HC, Kofler A, Nuesch R, Young J, Battegay M, Opravil M. Meta-analysis of randomized controlled trials of simplified versus continued protease inhibitor-based antiretroviral therapy in HIV-1-infected patients. AIDS. 2003 Nov 21;17(17):2451-9. doi: 10.1097/00002030-200311210-00007. PMID 14600516
- [Background] Drechsler H, Powderly WG. Switching effective antiretroviral therapy: a review. Clin Infect Dis. 2002 Nov 15;35(10):1219-30. doi: 10.1086/343050. Epub 2002 Oct 21. PMID 12410482
- [Background] Martinez E, Conget I, Lozano L, Casamitjana R, Gatell JM. Reversion of metabolic abnormalities after switching from HIV-1 protease inhibitors to nevirapine. AIDS. 1999 May 7;13(7):805-10. doi: 10.1097/00002030-199905070-00009. PMID 10357379
- [Background] Moyle G, Baldwin C, Mandalia S, Comitis S, Burn P, Gazzard B. Changes in metabolic parameters and body shape after replacement of protease inhibitor With efavirenz in virologically controlled HIV-1-positive persons: single-arm observational cohort. J Acquir Immune Defic Syndr. 2001 Dec 1;28(4):399-401. doi: 10.1097/00126334-200112010-00016. No abstract available. PMID 11707680
- [Derived] Lambert-Niclot S, Grude M, Meynard JL, Marcelin AG, Valantin MA, Flandre P, Izopet J, Moinot L, Bouteloup V, Calvez V, Katlama C, Girard PM, Morand-Joubert L. Ultrasensitive Human Immunodeficiency Virus Type 1 Viral Load as a Marker of Treatment Choice for Simplification Strategies. Clin Infect Dis. 2018 Nov 28;67(12):1883-1889. doi: 10.1093/cid/ciy382. PMID 29767684
- [Derived] Meynard JL, Bouteloup V, Landman R, Bonnard P, Baillat V, Cabie A, Kolta S, Izopet J, Taburet AM, Mercie P, Chene G, Girard PM; KALESOLO Study Group. Lopinavir/ritonavir monotherapy versus current treatment continuation for maintenance therapy of HIV-1 infection: the KALESOLO trial. J Antimicrob Chemother. 2010 Nov;65(11):2436-44. doi: 10.1093/jac/dkq327. Epub 2010 Sep 15. PMID 20843990
- See also: Click here for more information about this study: KALESOLO — http://www.imea.fr/